CLINICAL TRIAL: NCT00840515
Title: A Phase 2,Double Blind Randomized Study of PraevoSkin,a Melatonin Containing Emulsion, in the Prevention of Radiation Induced Dermatitis.
Brief Title: PraevoSkin Emulsion in the Prevention of Radiation Induced Dermatitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pharm Olam Pharmaceuticals Ltd. (Other)
Responsible Party: Roni Eilon, Pharm Olam Pharmaceutics Ltd.
Other Study IDs: SMC-5467; 20080772
Record Dates: First submitted 2009-02-07; First posted 2009-02-10 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Prevention of Radiation Induced Dermatitis.

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Emulsion

SUMMARY:
A phase 2 double blind randomised study of PraevoSkin,a melatonin containing emulsion, in the prevention of radiation induced dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients at least 18 years with unilateral breast cancer following lumpectomy +/- chemotherapy.
2. Planned to receive 50 Gy whole breast irradiation +/- boost to tumor bed.
3. ECOG PERFORMANCE STATUS 0-1.
4. Capable of giving written informed consent and following instructions for applying study emulsion or placebo as per control.
5. No co-morbidities known to affect radiotherapy reactions.
6. No co-existing acute or chronic skin disease.
7. No evidence of infection or inflammation of breast to be treated.
8. Not receiving chemotherapy during radiotherapy course.Biological therapy (e.g. Herceptin) or hormone therapy will be allowed during the study.

Exclusion Criteria:

1. Chemotherapy within 4 weeks prior to planned start of radiation or chemotherapy planned during radiation.
2. Prior radiotherapy to any site.
3. Collagen vascular disease.
4. Diabetes mellitus requiring medication.
5. Uncontrolled hypertension.
6. Participation in other clinical study.
7. Any contra-indicating to treatment with Melatonin.
8. History of allergy to peanuts or fragrances.
9. History of severe allergic reactions (e.g. asthma).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patientsplanned to receive whole breast radiation.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-06 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Digital Camera | Weekly